CLINICAL TRIAL: NCT06047470
Title: Macronutrients in Lactating NICU Parents - Impact of Kangaroo Care
Acronym: MILK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 1982835
Record Dates: First submitted 2023-08-01; First posted 2023-09-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Lactation Disorder With Baby Delivered; Nutrition Disorder, Infant
Keywords: Lactation; Kangaroo Care; NICU; Breast milk; Nutrition; Skin to skin
MeSH Terms: conditions — Infant Nutrition Disorders; Breast Feeding | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Intervention Model Description: This study is a mixed methods study comprising of a randomized, crossover interventional trial of Kangaroo Care vs Control and milk expression, study of implementation of scheduled Kangaroo Care in the UC Davis NICU, and qualitative interviews of providers and parents to understand their attitudes and experiences with Kangaroo Care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kangaroo Care Arm (KC) (Active Comparator): Lactating parents will be asked to arrive at the NICU 2 hours after they have fully expressed their breasts at home and to provide their infants with kangaroo care for 1 hour. Following KC and while still at the infant's bedside, lactating parents will be asked to pump from both of their breasts using a hospital grade pump available in the NICU. Study personnel will weigh the collected milk to determine the total volume of milk expressed by mass. The milk collected from both breasts will be gently swirled six times or more until the fat layer is incorporated in the bottle and will be combined into one bottle. Study personnel will take one 6 mL aliquot from the collected milk for compositional analysis. The remainder of the milk will be saved in the NICU per routine so that it can be fed to the infant later.
  Interventions: Behavioral: Kangaroo Care
- Control Arm (CON) (Placebo Comparator): Lactating parents will be asked to arrive at the NICU 3 hours after they have fully expressed their breasts at home. Lactating parents will be taken to a private room where they will be asked to pump from both of their breasts using a hospital grade pump available in the NICU. Study personnel will weigh the collected milk to determine the total volume of milk expressed by mass. The milk collected from both breasts will be gently swirled six times or more until the fat layer is incorporated in the bottle and will be combined into one bottle. Study personnel will take one 6 mL aliquot from the collected milk for compositional analysis. The remainder of the milk will be saved in the NICU per routine so that it can be fed to the infant later. Lactating parents will then provide their infants with kangaroo care for 1 hour.
  Interventions: Behavioral: No Kangaroo Care

INTERVENTIONS:
Behavioral: Kangaroo Care — Lactating parents will participate in kangaroo care (holding an infant upright, directly on the chest with skin-to-skin contact) prior to expressing a breast milk sample.
  Arms: Kangaroo Care Arm (KC)
Behavioral: No Kangaroo Care — Lactating parents will provide a breast milk sample after having no contact with their infant for at least 6 hours.
  Arms: Control Arm (CON)

SUMMARY:
The goal of this clinical trial is to learn about the impact of Kangaroo Care (holding your baby skin-to-skin on your chest) in lactating parents with babies in the Neonatal Intensive Care Unit (NICU) that cannot directly breastfeed.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn about the impact of Kangaroo Care (holding your baby skin-to-skin on your chest) in lactating parents with babies in the Neonatal Intensive Care Unit (NICU) that cannot directly breastfeed.

The main questions it aims to answer are:

* The impact on breast milk volume and macronutrient content (calories, fat, proteins, and carbohydrates)
* Parental experience and perceptions with Kangaroo Care in the University of California (UC) Davis NICU.

Parental participants will:

* Come to the UC Davis NICU for scheduled visits - 4 total visits in a 10 day period.
* Perform Kangaroo Care (holding your baby skin to skin on your chest) for one hour (nurses and other staff will help you place baby comfortably on your chest and be there to help with any questions/concerns while holding)
* Express breast milk per visit schedule (Either before or after Kangaroo Care) using hospital grade pump provided by the NICU
* Provide breast milk sample for analysis (6ml or just over a teaspoon)
* Participate in a brief interview over Zoom (no video required) - this will be about 20 minutes in length

Healthcare provider participants will:

•Participate in a brief interview over Zoom (no video required) - this will be about 20 minutes in length

ELIGIBILITY:
Inclusion Criteria:

Lactating Parent/Infant Dyads:

1. Lactating parents of infants who are currently admitted to the UCDMC NICU and are expected to remain in the NICU for at least 2 weeks from study enrollment
2. Lactating parent is 18 years of age or older
3. Infant with prematurity or other conditions prohibiting nutritive feeding at the breast during the study period
4. Lactating parent plans to feed their infants breast milk for at least 1 month
5. Lactating parent is willing to refrain from tandem feeding another child during the study period
6. Willing to refrain from enrolling infant in an interventional research study that may impact growth or feeding tolerance during the study period
7. Lactating parent is willing to use a hospital grade pump available in the NICU to express milk for sample collection
8. Lactating Parent that is willing to travel to UCDMC on 4 occasions within a 10 day period for study visits

Providers/staff:

1. Physicians, nurses, fellows, residents, and NICU staff involved in the implementation of Kangaroo care for the MILK study.

Exclusion Criteria:

1. Infant less than 1 week of age at enrollment
2. Lactating parents expressing breast milk for more than one infant
3. Lactating parents who are currently or plan to tandem feed another child during the study period
4. Lactating parents that are participating in an interventional research study that could influence breast milk production.
5. Lactating parents with infants deemed by primary investigator/primary care team to be too unstable for kangaroo care
6. Lactating parents that are unwilling to participate in kangaroo care
7. Dyads that have participated in nutritive feeding at the breast
8. Lactating parents that use recreational drugs that contraindicate breastfeeding/provision of breast milk
9. Lactating parents taking therapies, supplements, or medications that are incompatible with breastfeeding/provision of breast milk to their infant
10. Lactating parents using, or planning to use, any over-the-counter or prescription medication for the purpose of increasing milk supply (including domperidone, fenugreek, turmeric, blessed milk thistle, Brewer's yeast, or lactation cookies)
11. Lactating parents that are involuntarily confined
12. Lactating parents that are adults unable to consent
13. Lactating parents unwilling to travel to UC Davis NICU for study visits
14. Anyone deemed unfit for participation by the investigator(s)

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Breast milk calories (kcal/dL) by kangaroo care intervention | 10 days
  The difference in expressed breast milk caloric composition/energy content) between samples collected after participating in kangaroo care and those collected after having no contact with the infant for at least 6 hours.
Breast milk fat (g/dL) by kangaroo care intervention | 10 days
  The difference in expressed breast milk fat content between samples collected after participating in kangaroo care and those collected after having no contact with the infant for at least 6 hours.
Breast milk protein (g/dL) by kangaroo care intervention | 10 days
  The difference in expressed breast milk protein content between samples collected after participating in kangaroo care and those collected after having no contact with the infant for at least 6 hours.
Breast milk carbohydrate (g/dL) by kangaroo care intervention | 10 days
  The difference in expressed breast milk carbohydrate content between samples collected after participating in kangaroo care and those collected after having no contact with the infant for at least 6 hours.
Breast milk volume in mL by kangaroo care intervention | 10 days
  The difference in expressed breast milk volume expression between samples collected after participating in kangaroo care and after having no contact with the infant for at least 6 hours.
Implementation of scheduled Kangaroo Care Visits in the UC Davis NICU - KC time | 10 days
  Record minutes spent in Kangaroo Care during each study visit
Implementation of scheduled Kangaroo Care Visits in the UC Davis NICU - KC incomplete | 10 days
  Record reasons for KC visits lasting less than 60 minutes - including infant causes (clinical instability, intolerance, technical issues with equipment) and parental causes (parental discomfort/anxiety, parental scheduling conflict, need to use restroom/express breast milk)
Implementation of scheduled Kangaroo Care Visits in the UC Davis NICU - Parental attitudes | 9 months
  Qualitative survey (via zoom) of parents after study visit completion to better understand attitudes and experiences with scheduled Kangaroo Care visits.
Implementation of scheduled Kangaroo Care Visits in the UC Davis NICU - Provider attitudes | 9 months
  Qualitative survey (via zoom) of NICU providers after participation in study visit completion to better understand attitudes and experiences with scheduled Kangaroo Care visits.

SECONDARY OUTCOMES:
Duration of breast milk provision | 9 months
  Determine the length of time that breast milk is provided to the infant during the infant's hospital stay.
Infant growth (Birth weight and discharge weight in grams) during NICU hospitalization | 9 months
  Examine infant growth during NICU hospitalization, recording the birth weight and discharge weight
Infant growth (Birth length and discharge length in cm) during NICU hospitalization | 9 months
  Examine infant growth during NICU hospitalization, recording the birth weight and discharge weight
Infant growth (Birth head circumference and discharge head circumference in cm) during NICU hospitalization | 9 months
  Examine infant growth during NICU hospitalization, recording the birth weight and discharge weight
Infant growth (Birth weight z-score and discharge weight z-score) during NICU hospitalization | 9 months
  Examine infant growth during NICU hospitalization, recording the birth weight z-score and discharge weight z-score
Infant growth (Birth length z-score and discharge length z-score) during NICU hospitalization | 9 months
  Examine infant growth during NICU hospitalization, recording the birth weight z-score and discharge weight z-score
Infant growth (Birth head circumference z-score and discharge head circumference z-score) during NICU hospitalization | 9 months
  Examine infant growth during NICU hospitalization, recording the birth weight z-score and discharge weight z-score

CONTACTS AND LOCATIONS:
Overall Officials: Kara Kuhn-Riordon, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Section on Breastfeeding. Breastfeeding and the use of human milk. Pediatrics. 2012 Mar;129(3):e827-41. doi: 10.1542/peds.2011-3552. Epub 2012 Feb 27. PMID 22371471
- [Background] Lucas A, Cole TJ. Breast milk and neonatal necrotising enterocolitis. Lancet. 1990 Dec 22-29;336(8730):1519-23. doi: 10.1016/0140-6736(90)93304-8. PMID 1979363
- [Background] Sisk PM, Lovelady CA, Dillard RG, Gruber KJ, O'Shea TM. Early human milk feeding is associated with a lower risk of necrotizing enterocolitis in very low birth weight infants. J Perinatol. 2007 Jul;27(7):428-33. doi: 10.1038/sj.jp.7211758. Epub 2007 Apr 19. PMID 17443195
- [Background] Schanler RJ, Shulman RJ, Lau C. Feeding strategies for premature infants: beneficial outcomes of feeding fortified human milk versus preterm formula. Pediatrics. 1999 Jun;103(6 Pt 1):1150-7. doi: 10.1542/peds.103.6.1150. PMID 10353922
- [Background] Furman L, Taylor G, Minich N, Hack M. The effect of maternal milk on neonatal morbidity of very low-birth-weight infants. Arch Pediatr Adolesc Med. 2003 Jan;157(1):66-71. doi: 10.1001/archpedi.157.1.66. PMID 12517197
- [Background] Vohr BR, Poindexter BB, Dusick AM, McKinley LT, Higgins RD, Langer JC, Poole WK; National Institute of Child Health and Human Development National Research Network. Persistent beneficial effects of breast milk ingested in the neonatal intensive care unit on outcomes of extremely low birth weight infants at 30 months of age. Pediatrics. 2007 Oct;120(4):e953-9. doi: 10.1542/peds.2006-3227. PMID 17908750
- [Background] Vohr BR, Poindexter BB, Dusick AM, McKinley LT, Wright LL, Langer JC, Poole WK; NICHD Neonatal Research Network. Beneficial effects of breast milk in the neonatal intensive care unit on the developmental outcome of extremely low birth weight infants at 18 months of age. Pediatrics. 2006 Jul;118(1):e115-23. doi: 10.1542/peds.2005-2382. PMID 16818526
- [Background] Kumar RK, Singhal A, Vaidya U, Banerjee S, Anwar F, Rao S. Optimizing Nutrition in Preterm Low Birth Weight Infants-Consensus Summary. Front Nutr. 2017 May 26;4:20. doi: 10.3389/fnut.2017.00020. eCollection 2017. PMID 28603716
- [Background] Martin CR, Ling PR, Blackburn GL. Review of Infant Feeding: Key Features of Breast Milk and Infant Formula. Nutrients. 2016 May 11;8(5):279. doi: 10.3390/nu8050279. PMID 27187450
- [Background] Mimouni FB, Lubetzky R, Yochpaz S, Mandel D. Preterm Human Milk Macronutrient and Energy Composition: A Systematic Review and Meta-Analysis. Clin Perinatol. 2017 Mar;44(1):165-172. doi: 10.1016/j.clp.2016.11.010. PMID 28159203
- [Background] Acuna-Muga J, Ureta-Velasco N, de la Cruz-Bertolo J, Ballesteros-Lopez R, Sanchez-Martinez R, Miranda-Casabona E, Miguel-Trigoso A, Garcia-San Jose L, Pallas-Alonso C. Volume of milk obtained in relation to location and circumstances of expression in mothers of very low birth weight infants. J Hum Lact. 2014 Feb;30(1):41-6. doi: 10.1177/0890334413509140. Epub 2013 Nov 8. PMID 24212300
- [Background] Miles MS, Funk SG, Carlson J. Parental Stressor Scale: neonatal intensive care unit. Nurs Res. 1993 May-Jun;42(3):148-52. PMID 8506163
- [Background] Health WHOR, Organization WH, UNAIDS. Kangaroo Mother Care: A Practical Guide. World Health Organization; 2003.
- [Background] Hill PD, Aldag JC. Milk volume on day 4 and income predictive of lactation adequacy at 6 weeks of mothers of nonnursing preterm infants. J Perinat Neonatal Nurs. 2005 Jul-Sep;19(3):273-82. doi: 10.1097/00005237-200507000-00014. PMID 16106236
- [Background] Hill PD, Aldag JC, Chatterton RT. Effects of pumping style on milk production in mothers of non-nursing preterm infants. J Hum Lact. 1999 Sep;15(3):209-16. doi: 10.1177/089033449901500310. PMID 10578798
- [Background] Lau C, Hurst NM, Smith EO, Schanler RJ. Ethnic/racial diversity, maternal stress, lactation and very low birthweight infants. J Perinatol. 2007 Jul;27(7):399-408. doi: 10.1038/sj.jp.7211770. PMID 17592486
- [Background] Parker LA, Sullivan S, Krueger C, Kelechi T, Mueller M. Strategies to increase milk volume in mothers of VLBW infants. MCN Am J Matern Child Nurs. 2013 Nov-Dec;38(6):385-90. doi: 10.1097/NMC.0b013e3182a1fc2f. PMID 24145494
- [Background] Coskun D, Gunay U. The Effects of Kangaroo Care Applied by Turkish Mothers who Have Premature Babies and Cannot Breastfeed on Their Stress Levels and Amount of Milk Production. J Pediatr Nurs. 2020 Jan-Feb;50:e26-e32. doi: 10.1016/j.pedn.2019.09.028. Epub 2019 Oct 28. PMID 31672261